CLINICAL TRIAL: NCT05990101
Title: HYPoxaEmic Respiratory Failure and Awake Prone Ventilation
Acronym: Hyper-AP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/6-1517-981
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Respiratory Failure; Hypoxemia
Keywords: Awake prone; Respiratory failure; ARDS; Hypoxaemia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to the awake prone or standard care groups on a 1:1 ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: By the nature of the awake prone intervention, it will not be possible to blind clinicians; however, interventions will be blinded to data analysts and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP group (Experimental): Awake prone position (APP) for 4 or more hours per day in addition to standard care for the first 72 hours from randomisation. After the initial period, use of APP is at discretion of the treating clinician. Awake prone can be discontinued earlier if patients meets pre-specified criteria of sustained improvement.
  Interventions: Behavioral: Awake prone position (APP)
- Control group (No Intervention): Standard care excluding APP

INTERVENTIONS:
Behavioral: Awake prone position (APP) — Awake prone position for 4 or more hours per day for the first 72 hours following randomisation.
  Arms: APP group

SUMMARY:
The goal of this prospective multi-centre randomised controlled trial is to determine if addition of awake prone positioning to standard oxygen, high flow oxygen therapy and non-invasive ventilation may reduce the rates of endotracheal intubation and mechanical ventilation.

DETAILED DESCRIPTION:
Effectiveness of prone position in mechanically ventilated patients was investigated extensively. During the Covid-19 pandemic a sudden increase in cases of acute respiratory failure, resulted in renewed interest and numerous studies on applying this concept in spontaneously breathing patients and using this in conjunction with less invasive respiratory support. However, evidence form the Covid-19 trials may not be directly extrapolated to other acute respiratory distress causes (for example bacterial pneumonia) as pathology of lung injury is distinctly different. Even though first reports of awake prone positioning were published nearly 30 years ago, but to date there are no prospective randomised trials in adult population treated for acute lung injury unrelated to Covid-19. Existing publications range from case reports (lung transplantation and drowning cases) to small feasibility trials involving 15-20 patients and also neonatal and paediatric populations. Considering that patients with acute lung injury constitute a significant proportion of routine intensive care unit population, results of this study would be highly relevant for the daily practice in intensive care medicine.We are aiming to conduct a prospective multi-centre randomised controlled trial comparing standard care alone with awake prone positioning and standard care in spontaneously breathing patients admitted to Intensive or Intermediate Care Units for acute non-Covid-19 hypoxemic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to intensive care unit for acute hypoxemic respiratory failure.
* Acute hypoxemic respiratory failure is defined by respiratory rate ≥25 breaths/min, and partial pressure of oxygen in the arterial blood (PaO2)/fraction of inspired oxygen (FiO2) ≤300 mm Hg or oxygen saturation (SpO2)/fraction of inspired oxygen (FiO2) ratio <235 while spontaneously breathing under standard oxygen with oxygen flow rate of at least 10 L/min, high flow oxygen therapy or non-invasive ventilation. For patients under standard oxygen, FiO2 is calculated according to the following formula: FiO2=0.21 + 0.03 per litre of supplemental oxygen.
* Informed consent

Exclusion Criteria:

* impaired consciousness - Glasgow coma score <14;
* inability to cooperate or prone position intolerance;
* immediate indications for endotracheal intubation;
* patients with do-not-intubate order at time of inclusion;
* patients with contraindication to high flow oxygen therapy (HFOT) or non-invasive ventilation (NIV);
* Partial pressure of carbon dioxide (PaCO2) above 50 mm Hg and quantitative measure of the acidity (pH) <7,3;
* vasopressor dose >0.3 µg/kg/min of norepinephrine-equivalent to maintain systolic blood pressure >90 mmHg;
* Covid-19 positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of endotracheal intubation | Within 30 days of randomisation
  Incidence of endotracheal intubation in both groups

SECONDARY OUTCOMES:
Mortality | Within 1 year of randomisation
  Mortality during intensive care unit stay, in hospital, at day 90 and at 1 year
Duration of mechanical ventilation | Within 30 days of randomisation
  Total number of mechanical ventilation days from endotracheal intubation to discharge from intensive care unit
Length of intensive care unit and hospital stay | Within 30 days of randomisation
  Total cumulative number of days spent in intensive care unit and hospital
One year mortality | Within 1 year of randomisation
  Incidence or death during one year of randomisation
Health related quality of life | Within 1 year of randomisation
  Heath related quality of life assessed by Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) one year of randomisation

OTHER OUTCOMES:
Tolerance of awake prone positioning | Within 72 hours of randomisation
  Proportion of patients in the intervention group completing at least 4 hours per day of awake prone positioning and number of awake prone hours per day

CONTACTS AND LOCATIONS:
Overall Officials: Ieva Jovaisiene, Dr, Principal Investigator — Vilnius University Hospital Santaros Klinikos; Mandeep K Phull, Dr, Principal Investigator — Barking, Havering and Redbridge University Hospitals NHS Trust; Tomas Jovaisa, Prof, Principal Investigator — Vilnius University Hospital Santaros Klinikos
Locations (4):
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Republican Vilnius University Hospital, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Barking, Havering and Redbridge University Hospitals NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No